CLINICAL TRIAL: NCT05107518
Title: Turkish Version, Validity and Reliability Study of the "Children Participation Assessment Scale"
Brief Title: Children Participation Assessment Scale
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Rabia ZORLULAR, principal investigator, Gazi University
Other Study IDs: Children Participation
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Child Development; Physical Disability; Participation, Patient
Keywords: child development; children participation; validity; version
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Children Participation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- children with physical disabilities: his study was designed to examine the validity and reliability of the Turkish version of the Children Participation Assessment Scale. While examining the validity of the scale in children, it was planned to use the Child Health Questionnaire-(CSA) scale, which had previously been shown to be reliable and valid in healthy children with different disability levels.
  Interventions: Behavioral: Children Participation Assessment Scale

INTERVENTIONS:
Behavioral: Children Participation Assessment Scale — Evaluation is carried out to examine the validity and reliability of the Turkish version of the Children Participation Assessment Scale. While examining the validity of the scale in children, it was planned to use the Child Health Questionnaire scale, which had previously been shown to be reliable and valid in healthy children with different disability levels.
  Other Names: Child Health Questionnaire scale

SUMMARY:
Increasing the number of Turkish versions of questionnaires evaluating participation will increase the variety of assessment methods. This study aims to evaluate the Turkish version, validity and reliability of the Children Participation Assessment Scale.

DETAILED DESCRIPTION:
This study was designed to examine the validity and reliability of the Turkish version of the Children Participation Assessment Scale. Translation and cultural adaptation of the questionnaire will be designed according to an appropriate procedure. The original English version of the questionnaire is fluent in English; It will be translated into Turkish by two people, one a physiotherapist and the other a linguist. Translators will come together and combine the questionnaires translated into Turkish into a single translation. The questionnaire translated into Turkish will then be translated back into English by two sworn translators whose mother tongue is English and who know Turkish well. The questionnaire, which was translated from Turkish to English again, will be synthesized by the translation team and turned into a single translation and its compatibility with the original will be evaluated. 250 children between the ages of 6 and 12 with physical disabilities and their parents will be included in this study. Children and parents with serious visual and auditory problems and who do not volunteer to participate in the study will be excluded from the study. While examining the validity of the scale in children, it was planned to use the Child Health Questionnaire scale, which had previously been shown to be reliable and valid in healthy children with different disability levels. The questions in the data collection form will be asked to the parents in the form of face-to-face interviews.

ELIGIBILITY:
Inclusion Criteria:

* 6-12 years old
* physically disability
* adequate cognitive level

Exclusion Criteria:

* severe visual or auditory problems
* children and parents who did not volunteer to participate in the study

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 250 children aged 6-12 with physical disabilities and their parents will be included.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Children Participation Assessment Scale | 6-12 years
  Children Participation Assessment scale is an assessment tool that includes all work-occupation areas (daily life and activities, play, leisure time, social participation, work, sleep/rest). Children Participation Assessment Scale, used in children aged 6-12 It has two versions, child and parent version.

SECONDARY OUTCOMES:
Child Health Questionnaire | 5-18 years
  he Child Health Questionnaire (CHQ) is a generic health instrument designed to capture the physical and psychosocial well-being of children independently from the underlying disease.he purpose of the instrument is to evaluate the functional health and well-being of children aged 5-18 years via parent-proxy report.

CONTACTS AND LOCATIONS:
Overall Officials: rabia eraslan, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Amini M, Hassani Mehraban A, Rostamzadeh O, Mehdizadeh F. Psychometric Properties of the Iranian-Children Participation Questionnaire (I-CPQ) When Used with Parents of Preschool Children with Cerebral Palsy. Occup Ther Health Care. 2017 Oct;31(4):341-351. doi: 10.1080/07380577.2017.1382753. Epub 2017 Oct 17. PMID 29039716
- [Background] Amini M, Hassani Mehraban A, Pashmdarfard M, Cheraghifard M. Reliability and validity of the Children Participation Assessment Scale in Activities Outside of School-Parent version for children with physical disabilities. Aust Occup Ther J. 2019 Aug;66(4):482-489. doi: 10.1111/1440-1630.12569. Epub 2019 Jan 30. PMID 30697766
- [Background] Parsons SK, Shih MC, Mayer DK, Barlow SE, Supran SE, Levy SL, Greenfield S, Kaplan SH. Preliminary psychometric evaluation of the Child Health Ratings Inventory (CHRIs) and Disease-Specific Impairment Inventory-Hematopoietic Stem Cell Transplantation (DSII-HSCT) in parents and children. Qual Life Res. 2005 Aug;14(6):1613-25. doi: 10.1007/s11136-005-1004-2. PMID 16110940